CLINICAL TRIAL: NCT03201926
Title: Development and Clinical Application of Invalid Foods Using Mealworms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joon Seong Park, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3-2017-0077
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Pancreatobiliary Disease; Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mealworms (Experimental): mealworms
  Interventions: Dietary Supplement: mealworms
- grain powder (Placebo Comparator): grain powder
  Interventions: Dietary Supplement: grain powder

INTERVENTIONS:
Dietary Supplement: mealworms — 10g , 3 times a day , po, 2 months
  Arms: mealworms
Dietary Supplement: grain powder — grain powder, 10g ,3times one day,2months
  Arms: grain powder

SUMMARY:
Malnutrition in cancer patients continues after surgery and worsens the patient's overall health and quality of life. Previous studies reported edible insects in patients' diets increased postoperative muscle mass and weight gain. Therefore, by using nutritionally excellent mealworms for a long time, it is proved that nutritional status and survival rate are improved, leading to development of various products of edible insects.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery with pancreaticobiliary disease and liver cancer (metastatic liver cancer)
* Karnofsky performance status ≥ 70
* Patients who can communicate without difficulty in obtaining a consent form for the test

Exclusion Criteria: Patients with any of the following criteria are excluded.

* Patients who underwent palliative surgery
* Patients with uncontrolled pre-operative disease
* Previous history of surgery affecting nutritional status
* Pregnant and lactating women
* Patients with allergy to mealworms

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of Body mass index | Changes from baseline nutition index at Preoperative 1 day, Postoperative 14 days (one week after take mealworms), Postoperative 2 months( two months after take mealworms)
  Improvement of Nutrition index ( Body cell mass, Soft lean mass, Fat free mass, Fat mass)

SECONDARY OUTCOMES:
Improvement of Body weight change | Changes from baseline Body weight at Preoperative 1 day, Postoperative 14 days (one week after take mealworms), Postoperative 2 months( two months after take mealworms)
  weight in kilograms, height in meters, BMI in kg/m^2
Improvement of Immune Function Index | Changes from baseline nutition index at Preoperative 1 day, Postoperative 14 days (one week after take mealworms), Postoperative 2 months( two months after take mealworms)
  Improvement of Immune parameters(T cell, INF-r, TNF-a, NK cell, IL-1, IL-2)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HS, Lee YS, Jang SY, Jun SY, Lim JH, Kim IK, Kim HM, Park JS. Clinical application of invalid foods using mealworms and evaluation of nutrition status and immune function: a study protocol for a randomized, double blind, placebo-controlled trial. BMC Nutr. 2019 Nov 18;5:44. doi: 10.1186/s40795-019-0307-6. eCollection 2019. PMID 32153957